CLINICAL TRIAL: NCT07362732
Title: Exploratory Study on the Treatment of Recurrent and Refractory Hematological Malignancies With WGb-0302 Injection
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Professor, Sichuan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LNP-mRNA for BCMA
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WGb-0302 injection, Escalation doses (Experimental)
  Interventions: Drug: WGb-0302 injection
- WGb-0302 injection, Extended doses (Experimental)
  Interventions: Drug: WGb-0302 injection

INTERVENTIONS:
Drug: WGb-0302 injection — WGb-0303 injection

SUMMARY:
At present, the treatment of multiple myeloma (MM) has evolved from traditional chemotherapy to a comprehensive model that includes targeted drugs, immunotherapy, etc. However, the prognosis of recurrent/refractory MM patients remains severe. For patients who are already resistant to multiple major drugs such as proteasome inhibitors, immunomodulators, and CD38 monoclonal antibodies, the prognosis is particularly poor. B-cell maturation antigen (BCMA) plays a crucial role in regulating B cell proliferation and survival. BCMA is expressed in various hematological malignancies such as multiple myeloma and has become an important biomarker, promising therapeutic target, and research direction for these diseases.

The advent of COVID-19 vaccine has brought LNP mRNA technology into the public's view. After years of development, it not only shines brilliantly in COVID-19 vaccine, but also is widely used in the treatment and exploration of cancer, rare diseases and other fields. The core of LNP mRNA technology targeting BCMA is to encapsulate the mRNA encoding specific proteins (such as anti BCMA related proteins) in lipid nanoparticles and deliver them to the body through intravenous or intramuscular injection. The experimental drug WGb 0302 injection is a BCMA based messenger RNA (mRNA) therapeutic drug, formed by loading mRNA encoding BCMA receptor related proteins onto lipid nanoparticles (LNP).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range: 18-75 years old, gender not limited;
* 2. Expected survival time exceeds 12 weeks;
* 3. According to the diagnostic criteria of the International Myeloma Working Group (IMWG) for multiple myeloma, the diagnosis is multiple myeloma (MM), and the expression of BCMA target antigen is confirmed by flow cytometry, bone marrow pathology, and immunohistochemistry.
* 4. Having measurable multiple myeloma lesions:
* 5. The physical fitness status score of the Eastern Cancer Collaboration Group (ECOG) is 0 or 1 point;
* 6. Before screening (at baseline), corresponding conditions should be met;
* 7. Male and female patients of appropriate age must use reliable methods of contraception before entering the trial, during the research process until 30 days after discontinuation of medication; Reliable contraceptive methods will be determined by the primary researchers or designated personnel;
* 8. Those who can understand this experiment and have signed the informed consent form.

Exclusion Criteria:

* 1. Accompanied by other uncontrolled malignant tumors;
* 2. Previously received chimeric antigen receptor therapy or other transgenic T cell therapy less than 6 months after the first administration;
* 3. Have received any anti myeloma treatment (including but not limited to chemotherapy, targeted therapy, immunotherapy, radiation therapy [excluding local radiotherapy for pain control], etc.) within 14 days prior to the first use of medication;
* 4. Known history of HIV or hepatitis B (HBsAg positive and HBV DNA reaching the detection limit) or hepatitis C virus (anti HCV positive) infection;
* 5. Participants with a history of CNS lymphoma, malignant cells in cerebrospinal fluid, or brain metastases;
* 6. Within 14 days prior to enrollment, there is an uncontrolled active infection. Note: If there is no evidence of active infection within 72 hours before enrollment, subjects who continue to use prophylactic antibiotics, antifungal drugs, or antiviral drugs are allowed;
* 7. Emergency treatment is required due to the impact of tumor masses, such as intestinal obstruction or vascular compression;
* 8. Suffering from serious diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage, poorly controlled hypertension, or other uncontrolled active diseases that hinder participation in the trial;
* 9. Unstable pulmonary embolism, deep vein thrombosis, or other significant arterial/venous thromboembolism events occurred within 30 days prior to enrollment. If receiving anticoagulant therapy, the treatment dose of participants must reach a stable level before enrollment;
* 10. Long term use of immunosuppressants due to autoimmune diseases or organ transplantation, except for recent or current inhaled corticosteroid therapy;
* 11. Any pregnant or breastfeeding woman, or participant who plans to conceive during or within 18 months after treatment;
* 12. The researcher believes that there are any other factors that are not suitable for the study participants to enter this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicity (DLT) | Within 90 days after the initial treatment
Maximum tolerated dose (MTD)or optimal biological dose (OBD) | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 2 years
Progression free survival (PFS) | From date of initial treatment until the date of first comfired progression or date of death from any cause, whichever came first, assessed up to 24 months